CLINICAL TRIAL: NCT06278363
Title: The Role of Sexual Nursing Care in Managing Sexual Dysfunctions in Stroke Patients
Brief Title: Sexual Nursing Care in Stroke Patients
Acronym: StrokeSex_23
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, co-investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: StrokeSex_23
Record Dates: First submitted 2024-02-09; First posted 2024-02-26 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Stroke
Keywords: Sexual nursing care; sexuality; Sexual health; sexual dysfunction; Stroke
MeSH Terms: conditions — Stroke; Sexuality; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: We aim to assess the effectiveness of an intervention in stroke subjects to increase awareness of sexual health, effectively manage sexual dysfunctions, reduce their frequency, and enhance psychophysical well-being.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant Masking: Participants are unaware of the treatment they are receiving. This helps prevent biases in reporting outcomes based on knowledge of the treatment.
  Care Provider Masking: The individuals providing care, such as therapists or nurses, are also unaware of the treatment assigned to each participant. This prevents them from inadvertently influencing outcomes based on their knowledge of the treatment.
  Investigator Masking: The individuals responsible for collecting and analyzing the data are blinded to the treatment allocation. This helps ensure impartiality and prevents biases in data interpretation.
  Outcomes Assessor Masking: Individuals responsible for assessing the outcomes of the study, such as evaluating patient progress or interpreting test results, are blinded to the treatment group to which participants belong. This prevents biases in outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sexual Nursing Care (Experimental): Group 1 patients receive "Sexual Nursing Care," involving personalized counseling by a nurse to address sexual dysfunctions post-stroke. The intervention includes partner involvement to foster new intimacy, sexual education, and exercises. Four 45-minute outpatient sessions with the nurse and partner are provided. Any emerging issues requiring diagnostic investigation will be communicated to the referring specialist.
  Interventions: Other: Sexual Nursing care
- Standard Nursing Care: (Active Comparator): Patients in Group 2 receive a standard nursing care approach. In this group, no specific structured interventions for sexual dysfunctions are provided. Management of sexual dysfunctions occurs based on the clinical case and standard care approach.
  Care sessions follow a routine program, without specific interventions for the sexual sphere.
  As in Group 1, any emerging issues during treatment that require further diagnostic investigation will be communicated to the referring specialist.
  Both groups will be evaluated for the impact of treatment not only quantitatively, through the analysis of the effect of counseling on sexual and relational aspects but also qualitatively, to investigate psychorelational changes and mood impact on the quality of life of the involved couples.
  Interventions: Other: Standard Nursing Care

INTERVENTIONS:
Other: Sexual Nursing care — The Sexual Nursing Care approach is a specialized intervention for stroke patients and partners, addressing sexual health needs. It includes personalized counseling sessions with trained nurses, assessing dysfunctions and medical history. Active partner involvement fosters intimacy and understanding. Both receive sexual education covering anatomy, physiology, and post-stroke changes. Recommendations for activities like Kegel exercises are provided. Structured outpatient sessions occur, lasting 45 minutes, facilitated by a nurse. Pre- and post-treatment assessments are conducted to identify contraindications. Emerging issues during treatment are promptly communicated for management. Sexual Nursing Care aims to holistically address post-stroke sexual health and relational needs, improving awareness and communication.
  Coaching and Counselling can be provided also via telemedicine.
  Arms: Sexual Nursing Care
Other: Standard Nursing Care — Group 2 patients receive standard nursing care without structured interventions for sexual dysfunctions. Management relies on clinical case and routine care procedures. No specific sexual sphere interventions are provided. Any emerging issues needing diagnostic investigation are reported to the specialist. Both groups are assessed quantitatively for counseling effects on sexual and relational aspects and qualitatively for psychorelational changes and mood impact on couple's quality of life.
  Arms: Standard Nursing Care:

SUMMARY:
The study aims to assess the impact of "sexual nursing care" on sexual dysfunctions in Italian stroke patients.

The method involves a randomized clinical trial with two groups: one receiving specific sexual care and the other standard care, both involving the partner. Various assessment scales are used, and four outpatient interventions are administered over six months.

Results indicate improvement in body awareness, management of sexual dysfunctions, relational dynamics, and quality of life for both patients and partners.

In conclusion, the importance of sexual health in stroke patients is highlighted as an indicator of quality of life. Targeted nursing interventions can facilitate timely diagnosis and a personalized approach to patients and partners.

DETAILED DESCRIPTION:
Introduction:

Stroke is a leading cause of disability in adults worldwide, affecting approximately 1.9-4.3% of individuals aged over 20. Patients often experience motor and cognitive issues post-stroke, with around 40% affected within a year. Moreover, sexual dysfunctions affect approximately 50% of stroke survivors, including erectile dysfunction and altered lubrication, impacting relationships and quality of life for both patients and caregivers.

Sexuality plays a significant role in an individual's overall well-being, yet the sexual health needs of stroke patients are often overlooked in clinical practice. This study aims to assess the role of sexual nursing care in addressing sexual dysfunctions among Italian stroke patients and improving overall psychophysical well-being.

Objectives of the Study:

The primary objective is to evaluate the effectiveness of sexual nursing care in enhancing sexual awareness, managing sexual dysfunctions, and improving overall psychophysical well-being among stroke patients. Secondary objectives include assessing improvements in psychorelational dynamics within couples and evaluating the benefits of nursing counseling on patients' and partners' quality of life.

Study Population:

The study will include patients with ischemic and hemorrhagic stroke admitted to the Physical Medicine and Rehabilitation Unit of AOU Policlinico "G. Martino" in Messina, Italy, during the subacute phase (1-3 months post-event).

Inclusion criteria: Clinical and neuroradiological diagnosis of stroke, aged 18-70 years.

Exclusion criteria: Pre-existing neurodegenerative diseases, endocrine-metabolic and psychiatric conditions interfering with sexual function, global aphasia, or other cognitive impairments hindering active participation.

Study Design and Procedures:

The study will employ a randomized clinical trial (RCT) design with block randomization. Patients will be allocated into two groups: Group 1 (GS) receiving sexual nursing care and Group 2 (GC) receiving standard nursing care. Both groups will involve the partner.

Before enrollment, patients will undergo a comprehensive assessment to identify contraindications and ensure adherence to exclusion criteria.

Sexual nursing care interventions will include counseling, sexual education, and exercises for sexual function improvement. Four outpatient interventions will be conducted bimonthly, each lasting 45 minutes and involving the nurse, patient, and partner.

The study will utilize a mixed-method approach, combining a quantitative assessment of counseling effects on sexual-relational aspects with a qualitative investigation into psychoemotional changes and mood disorders impacting the quality of life in stroke-affected couples.

Outcome Measures:

A battery of tests will be administered at baseline (T0), 3 months (T1), and 6 months (T2) to evaluate outcomes. Trained nurses, blinded to patient groupings, will conduct clinical scale assessments.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and neuroradiological diagnosis of ischemic or hemorrhagic stroke.
* Age between 18 and 70 years.
* Patients in the subacute phase (1-3 months post-event).

Exclusion Criteria:

* Pre-existing neurodegenerative diseases (e.g., multiple sclerosis).
* Endocrine-metabolic and psychiatric pathologies that may interfere with sexual function.
* Global aphasia or other cognitive impairments that hinder active participation in training.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of "sexual nursing care" intervention in enhancing sexual awareness | Patients are enrolled approximately one month after hospitalization following a stroke. They undergo bi-monthly outpatient sessions, indicating a continuous and structured treatment regimen.
  The "sexual nursing care" intervention involves personalized counseling by trained nurses, partner involvement, sexual education, and guidance for improving sexual function.
  The primary outcome assesses the impact on increasing sexual health awareness in stroke patients and partners. Evaluation includes a semi-structured interview for sexual dysfunctions, Female Sexual Function Index (FSFI) for women, and International Index of Erectile Function (IIEF) for men.

SECONDARY OUTCOMES:
psychosocial well-being and relational dynamics of stroke patients and their partners | Patients are enrolled approximately one month after hospitalization following a stroke. They undergo bi-monthly outpatient sessions, indicating a continuous and structured treatment regimen.
  The secondary aim is to assess the broader effects of "sexual nursing care" on the:
  1. psychosocial well-being and
  2. relational dynamics of stroke patients and partners. Through tailored counseling and interventions, the investigators aim to improve the couple's dynamics and overall quality of life.
  Outcome measures include:
  1. the Dyadic Adjustment Scale (DAS) for relational satisfaction
  2. the WHOQOL-Brief Scale to monitor quality of life changes By evaluating these objectives, the investigators aim to understand the broader impacts of "sexual nursing care," contributing to enhanced psychosocial well-being and relationships in stroke patients and partners.

CONTACTS AND LOCATIONS:
Overall Officials: Provvidenza Tommasello, MsC, Principal Investigator — IRCCS Centro Neurolesi Bonino Pulejo
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Italy/Messina, Italy

IPD SHARING:
Plan to Share IPD: No
We are considering the use of a cloud database to share anonymized patient data with other researchers, which would involve making individual participant data (IPD) available.

REFERENCES:
- [Result] Calabro RS, Manuli A. Sexual Function and Disability in the Neurorehabilitation Setting: An Urgent Need for a Multidisciplinary Approach. Innov Clin Neurosci. 2021 Oct-Dec;18(10-12):26-27. PMID 35096479
- [Result] Na Y, Htwe M, Rehman CA, Palmer T, Munshi S. Sexual dysfunction after stroke-A biopsychosocial perspective. Int J Clin Pract. 2020 Jul;74(7):e13496. doi: 10.1111/ijcp.13496. Epub 2020 Mar 5. PMID 32100415